CLINICAL TRIAL: NCT01385865
Title: Effect of Mulberry Leaf Extract on Blood Glucose in Subjects With Impaired Fasting Glucose
Brief Title: Effect of Mulberry Leaf Extract on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Collaborators: CHA University (Other); Ministry of Knowledge Economy, Korea (Unknown)
Responsible Party: Principal Investigator, Oran Kwon, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MLE_Biofood_2
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Morus alba

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mulberry leaf extract (Experimental)
  Interventions: Dietary Supplement: Mulberry leaf extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mulberry leaf extract — 18 tablets/day (6 tablets/serving x 3servings/day, mulberry leaf extract 336mg/1 tablet (800mg), 1-Deoxynojirimycin 4.3mg/1 g mulberry leaf extract), Duration: 4 weeks
  Arms: Mulberry leaf extract
Dietary Supplement: Placebo — 18 tablets/day (6 tablets/serving x 3servings/day, lactose 511mg/1 tablet (650mg)), Duration: 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of mulberry leaf extract on blood glucose in subjects with impaired fasting glucose.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of mulberry leaf extract on blood glucose in subjects with impaired fasting glucose. After 2 weeks run-in period for wash-out, subjects will randomly assigned to two groups, i.e. control group (placebo) or mulberry leaf extract group. They will intake placebo or mulberry leaf extract for 4 weeks. Biomarkers will be analyzed in blood samples in 0 and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 20 years
* Fasting glucose: 100mg/dl ≤ ~ ≤ 125mg/dl
* HbA1c: < 6.5%

Exclusion Criteria:

* Subject who has taken medicines, Chinese medicines and Health/Functional Foods which can affect glucose metabolism in 30 days prior to screening visit
* Subject who has taken part in other clinical trials in 30 days prior to screening visit
* Subject who is pregnant or breast feeding
* Subject who lost body weight over 4 kg in 30 days prior to screening visit
* Alcoholic
* Heavy smoker (≥ 20 cigarettes/day)
* Subject who has heart failure, coronary artery disease, uncontrolled hypertension (≥ 140/90mmHg), diabetes (fasting blood glucose ≥ 126mg/dL), renal dysfunction, liver failure, hyperthyroidism, hypothyroidism, cancer or mental disease
* Subject who has an allergy to the ingredients of study product

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose change with meal tolerance test | 0wk

SECONDARY OUTCOMES:
Blood glucose change with meal tolerance test | 4wk
Insulin and C-peptide changes with meal tolerance test | 0, 4 wk
Fasting blood glucose | 0, 4 wk
Insulin | 0, 4wk
C-peptide | 0, 4wk
Glycated albumin | 0, 4wk
High sensitivity C-reactive protein | 0, 4wk
Oxidized low-density lipoprotein | 0, 4wk
Malondialdehyde | 0, 4wk
Lipid profile (triglyceride, total cholesterol, low-density lipoprotein cholesterol, very-low-density lipoprotein cholesterol, high-density lipoprotein cholesterol) | 0, 4wk

CONTACTS AND LOCATIONS:
Overall Officials: Oran Kwon, Ph.D, Principal Investigator — Ewha Womans University; Sung Won Kwon, MD, Principal Investigator — CHA University; Seok Won Park, MD, Principal Investigator — CHA University; Moon Jong Kim, MD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea